CLINICAL TRIAL: NCT07162454
Title: A Triple-Blind Randomised Clinical Trial on the Effectiveness of CBD for Neuropathic Pain in Diabetic Foot Neuropathy
Brief Title: Effectiveness of CBD for Neuropathic Pain in Diabetic Foot Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, María del Sol Tejeda Ramírez, Podiatrist. Specialist in diabetic foot., Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24/193-EC_X
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Xerosis Cutis; Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Keywords: Diabetes mellitus; Diabetic foot; Diabetic neuropathy; Neuropathic pain; Cannabidiol; Urea 10%
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Diabetic Neuropathies; Neuralgia | interventions — Urea; Food, Formulated

STUDY DESIGN:
Intervention Model Description: Three groups were created and each group was assigned a different composition. A baseline and a final evaluation was performed after one month to assess the neuropathic pain and skin quality of the participants.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1. Complete formula. (Experimental): Participants in this group received a cream with cannabidiol, urea 10%, arnica and menthol as active ingredients during 1 month.
  Interventions: Drug: Group 1. Complete formula
- Group 2. Cannabidiol and Urea 10% formula. (Experimental): Participants in this group received a cream with cannabidiol, urea 10% as active ingredients during 1 month.
  Interventions: Drug: Group 2. Cannabidiol and Urea 10% formula.
- Group 3. Base formula. (Placebo Comparator): Participants in this group received a base cream with no active ingredients.
  Interventions: Drug: Group 3. Placebo formula.

INTERVENTIONS:
Drug: Group 1. Complete formula — After fulfilling the criteria and agreeing to participate in the study, patients who were included in group 1 after randomisation were evaluated and received a topical cream with cannabidiol, Urea 10%, arnica and menthol as active ingredients. After one month of application of the formula, a second evaluation was carried out.
  Arms: Group 1. Complete formula.
Drug: Group 2. Cannabidiol and Urea 10% formula. — After meeting the criteria and agreeing to participate in the study, the patients who were included in group 2 after randomisation were evaluated and received a topical cream containing cannabidiol and 10% urea. After one month of application of the formula, a second evaluation was carried out.
  Arms: Group 2. Cannabidiol and Urea 10% formula.
Drug: Group 3. Placebo formula. — Participants included in this group after randomisation received a formulation with no active ingredients included in its composition and were assessed at baseline and after one month.
  Arms: Group 3. Base formula.

SUMMARY:
Evaluation of cannabidiol and urea 10%.

DETAILED DESCRIPTION:
This study evaluated the impact of cannabidiol on neuropathic pain and the action of urea 10% on skin quality in patients with diabetic foot syndrome and diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients all biological sexes
* Patients of legal age (18 years).
* Patients without cognitive impairment
* Patients Diagnosed with diabetic neuropathy,
* Patients who were able to complete the neuropathic pain scale autonomously, cooperatively and independently.

Exclusion Criteria:

* Patients who declined participation
* Patients with critical ischaemia and
* Patients with a history of allergy or hypersensitivity to any of the components of the cream were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of neuropathic pain. | From randomisation and delivery of the assigned formula until the end of the intervention after one month of application.
  Neuropathic pain was assessed using the validated neuropathic pain assessment scale.

SECONDARY OUTCOMES:
Skin quality assessment | From randomisation and delivery of the assigned formula until the end of the intervention after one month of application.
  The assessment of skin quality was carried out using the validated questionnaire 'Injury Risk and Skin Quality Assessment Questionnaire'.

CONTACTS AND LOCATIONS:
Overall Officials: José Luis Lázaro Martinez, Podiatrist, Study Director — Clínica Universitaria de podología de la Universidad Complutense de Madrid
Locations (1):
- Facultad de Enfermería, Fisioterapia y Podología de la Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu DH, Cullen BD, Tang M, Fang Y. The Effectiveness of Topical Cannabidiol Oil in Symptomatic Relief of Peripheral Neuropathy of the Lower Extremities. Curr Pharm Biotechnol. 2020;21(5):390-402. doi: 10.2174/1389201020666191202111534. PMID 31793418
- See also: Research background on the effect of topical cannabidiol on various neuropathies. — https://pubmed.ncbi.nlm.nih.gov/31793418/